CLINICAL TRIAL: NCT02745886
Title: Chronic Metformin Treatment Induces a Dietary Restriction-like State in Overweight Human
Brief Title: Metformin Induces a Dietary Restriction-like State in Human
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wze2016009
Record Dates: First submitted 2016-04-01; First posted 2016-04-20 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Overweight Subjects; Metformin; Aging
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metformin group (Experimental): Metformin 0.85 twice daily for 6 months
  Interventions: Drug: metformin 0.85 twice daily for 6 months
- Standard diet group (No Intervention)
- CR group (Other): Calorie restriction diet will be given to this group.
  Interventions: Behavioral: Calorie restriction

INTERVENTIONS:
Drug: metformin 0.85 twice daily for 6 months
  Arms: Metformin group
Behavioral: Calorie restriction
  Arms: CR group

SUMMARY:
The fact that metformin treatment has been associated with reduced risk of cancer and cardiovascular disease raises the possibility of a beneficial role of metformin for other age-related diseases. The actions of metformin resemble the effects of calorie restriction (CR) to some extent, and microarray analyses have shown that metformin induces a gene expression profile that aligns with that of CR in animal. The aim of the study is to investigate whether metformin treatment can induce dietary restriction-like state in human.

Sixty overweight subjects will be included in this study, and participants will be divided 3 groups (20 cases in each group)including metformin group (0.85, twice daily), standard diet group, and CR group. All subjects will be treated 6 months. At the end of this study, blood samples and muscle samples will be obtained.

DETAILED DESCRIPTION:
Blood samples will be obtained from all individuals. blood lipids, inflammation markers, insulin, glucose, leptin,adiponectin, ala aminotransferase, asp aminotransferase, creatine phosphokinase,lactate dehydrogenase, alkaline phosphatase,bilirubin, cyclo-oxygenase, citrate synthase, renal function, leukocyte telomere length ratio, and telomerase activity will be measured before and after the treatments.Also, hyperinsulinemic-euglycemic clamp will be performed before and after the treatments. Muscle samples will be obtained by biopsy for 9 individuals (3 cases from each group) at the end of the study. Microarray analysis will be performed for the gene expression profile from the muscle samples. Other protein expressions such asadenosine monophosphate-activated protein kinase (AMPK), peroxisome proliferator-activated receptor coactivator 1a (PGC-1a) activity,will be checked by Western blot.

ELIGIBILITY:
Inclusion Criteria:

* Overweight
* Male

Exclusion Criteria:

* Female
* Obesity
* Using any other drugs
* < 18 years old
* > 60 years old
* Mental disorders
* Surgery history for abdomen

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The differences of gene expression profile among 3 groups. | 6 months
  The gene expression profile will be checked by microarray, and compared the number differences of pathways among 3 groups.

SECONDARY OUTCOMES:
The differences of insulin sensitivity in 3 groups | 6 months
  The insulin sensitivity will be measured by insulin clamp assays, and be compared before and after 6 months as well as among 3 group at the end of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Guangda Xiang, MD,PhD, Study Chair — Wuhan General Hospital
Locations (1):
- Zhang Jiajia, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes